CLINICAL TRIAL: NCT02909959
Title: A Phase II, Randomized, Double-blind, Placebo-controlled Study of Myrosinase-enriched Glucoraphanin, a Sulforaphane Precursor System, in Autism Spectrum Disorder
Brief Title: Sulforaphane for the Treatment of Young Men With Autism Spectrum Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-2059; 5KL2TR001109-05 (NIH)
Record Dates: First submitted 2016-09-07; First posted 2016-09-21 (Estimated); Results first posted 2020-05-15 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2019-06

CONDITIONS: Autism Spectrum Disorder; Autistic Disorder; Neurodevelopmental Disorder; Childhood Developmental Disorders, Pervasive
Keywords: sulforaphane; glucoraphanin; physiologic effects of drugs
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Neurodevelopmental Disorders | interventions — sulforaphane; glucoraphanin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sulforaphane (Active Comparator): Participants will take a sulforaphane supplement 3-8 tablets daily, with dose depending upon body weight. Each tablet contains 125 mg broccoli seed powder and 50 mg broccoli sprout extract, providing approximately 15 µmol sulforaphane.
  The weight-based dosing schedule is as follows:
  3 tablets (approx. 46.5 µmol SF) if <100 lb; 5 tablets (approx. 77.5 µmol SF) if 100-125 lb; 6 tablets (approx. 93 µmol SF) if 126-175 lb; 7 tablets (approx. 108.5 µmol SF) if 176-199 lb; 8 tablets (approx. 124 µmol SF) if ≥ 200 lb
  Interventions: Drug: Sulforaphane
- Placebo (Placebo Comparator): Participants in this arm will take placebo tablets that are identical in shape, size, and color to the sulforaphane tablets. The number of tablets taken per day corresponds to the weight-based schedule described for the sulforaphane arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sulforaphane — The investigational medicinal product is an uncoated tablet containing both glucoraphanin and myrosinase, the enzyme that converts glucoraphanin to sulforaphane in vivo. Participants in this arm will take 3-8 tablets by mouth once daily (dose depending upon weight) for 12 weeks.
  Other Names: Avmacol; glucoraphanin
  Arms: Sulforaphane
Drug: Placebo — Placebo tablets are uncoated and matched in appearance to the investigational medicinal product, containing inert components. Participants in this arm will take 3-8 tablets by mouth once daily (dose depending upon weight) for 12 weeks.
  Other Names: Control
  Arms: Placebo

SUMMARY:
The aim of this randomized controlled trial is to determine if a nutritional supplement containing broccoli sprout and seed extracts, a rich source of sulforaphane, is effective in reducing core symptoms of autism spectrum disorder (ASD). The study will also explore the safety and tolerability of a sulforaphane supplement in young men with ASD, as well as its effects on challenging neuropsychiatric symptoms that are commonly associated with ASD, such as hyperactivity, irritability, and repetitive movements.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a neurodevelopmental disorder affecting 1 in 68 children, including 1 in 42 boys, characterized by marked social communication impairment and restricted, repetitive behaviors and interests. Evidence-based pharmacological treatments available for the treatment of the defining symptoms of ASD are currently lacking.

While the etiology of ASD is not fully understood, the pathogenesis is hypothesized to involve cellular dysfunction, including increased oxidative stress, aberrant neuroinflammation, and reduced mitochondrial capacity, leading to synaptic dysfunction in at least a subset of individuals. Sulforaphane is a powerful upregulator of antioxidant response elements and heat shock proteins, which may lead to improved redox capacity, decreased inflammation, and improved mitochondrial functioning in individuals with ASD. A trial by Singh and colleagues (2014) provided preliminary evidence suggesting that sulforaphane derived from broccoli sprout extract can have beneficial effects for improving symptoms of autism.

In this study, young men ages 13-30 years old with moderate to severe autism spectrum disorder will be randomly assigned to receive either a sulforaphane supplement or placebo for a 12 week treatment treatment period, followed by a 4 week blinded discontinuation phase. The uncoated tablets each contain 125 mg broccoli seed extract and 50 mg broccoli sprout extract, corresponding to approximately 15 µmol sulforaphane per tablet. The dose will vary from 3-8 tablets daily depending upon the participant's weight. Matched placebo tablets contain only inert ingredients

A serum sample will be collected prior to starting treatment and at the end of the treatment phase to quantify sulforaphane metabolites. Clinical response will be assessed through clinician- and caregiver-rated measures of autism symptoms (Social Responsiveness Scale-2; Repetitive Behavior Scale- Revised), challenging symptoms commonly observed in individuals with developmental disabilities (Aberrant Behavior Checklist), and global severity of symptoms and improvement (Clinical Global Impression Scale). A blood sample will be collected at baseline and at the end of the treatment phase to check safety labs, and a saliva sample will be collected at baseline for a future study of genetic biomarkers associated with treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Males between ages 13-30 (inclusive) at the time of the consent
* Primary diagnosis of Autism Spectrum Disorder (ASD), confirmed by Diagnostic and Statistical Manual-5 (DSM-5) criteria and meeting the autism cut-off score of 9 or greater on the Autism Diagnostic Observation Schedule-2 (ADOS-2)
* Participant is capable of giving written informed consent or has a legally authorized representative (LAR) with sufficient capacity to provide written informed consent on the participant's behalf.
* Participant has a reliable informant (parent or caregiver) who has sufficient past and current knowledge of the subject and will oversee the administration of study medication and accompany the subject to each study visit.
* Participant and caregiver have reliable means of transportation to attend study visits.

Exclusion Criteria:

* Chronic medical illness that is not stable or would pose a risk to the participant if he participates in the trial
* History of clinical seizures within the 12 months preceding study enrollment
* Known genetic disorder that is presumed to be the cause of autism spectrum disorder (eg., Fragile x syndrome, tuberous sclerosis)
* Changes to psychopharmacological medications (e.g., stimulants, antidepressants, anxiolytics, antipsychotics) in the 4 weeks preceding study enrollment
* Significant changes to non-pharmacological treatments for ASD in the 4 weeks preceding study enrollment
* Chronic treatment with anti-inflammatory agents (e.g., ibuprofen, NSAIDs, corticosteroids)
* Clinically significant laboratory abnormalities at Screening visit (e.g., AST/ALT> two times the upper normal limits; serum creatinine > 1.2 mg/dl, TSH outside normal limits)
* Clinically significant findings on physical examination that investigator determines could increase risk of harm from participating in the study
* Participated in another clinical interventional trial or received an investigational product in the 30 days preceding study enrollment
* Previous therapeutic trial of sulforaphane or participation in a clinical trial in which sulforaphane was the investigational agent

Ages: 13 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Politte, M.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Carolina Institute for Developmental Disabilities, University of North Carolina School of Medicine, Carrboro, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to publish the results of this trial in a peer-reviewed journal and on ClinicalTrials.gov upon completion of the study. No personal identifiable participant data will be included in the reporting of results.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sulforaphane | Placebo
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sulforaphane | Placebo | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 15 | 31
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.8 (3.9) | 17.7 (4.1) | 17.2 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 24 | 24 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 23 | 22 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 19 | 21 | 40
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Social Responsiveness Scale-2 (SRS-2) Total Score at Baseline
Description: The Social Responsiveness Scale-2 (SRS-2) is a 65-item caregiver report that includes 5 subscales covering core symptom domains of ASD (Social Awareness, Social Cognition, Social Communication, Social Motivation, and Restricted Interests/ Repetitive Behaviors). The SRS-2 provides a T-score that is scaled such that the mean is 50 and the SD is 10. Higher scores indicate a higher presence and severity of autistic social impairment. A T-score of 76 or higher is considered "severe". T-scores between 66 and 75 are considered as "moderate". T-scores between 60 and 65 are considered "mild". A T-score below 60 is considered typical. The theoretical range of a T-score is 10 to 90. The actual range of the SRS-2 in this study is 45 to 90.
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
T-score | 75.6 (7.4) | 72.6 (4.6)
Statistical Analysis 1: Comparison: Sulforaphane vs Placebo; The null hypothesis is that the least-square mean of sulforaphane's SRS-2 T-score minus the least-square mean of placebo group's T-score is 0; Test type: Equivalence — Statistical significance was measured at the 0.05 alpha level for a two-sided test, so the rejection region for a normally distributed T-score was +/-1.96*SE(Diff), where SE(Diff) is the estimated standard error of the difference between the LS mean of sulforaphane and LS mean of the placebo group; p = 0.331, Mixed Models Analysis — The test was considered statistically significant if the p-value < 0.05; Mixed-effects model with random intercept and unstructured covariance matrix from baseline to week 16; Mean Difference (Final Values) = 2.96, Standard Error of Mean 3.03 — This analysis compares LS Mean Sulforaphane - LS Mean Placebo

2. Primary Outcome: Social Responsiveness Scale-2 (SRS-2) Total Score at Week 4
Description: as for outcome 1
Time Frame: Week 4
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
T-score | 74.1 (7.4) | 74.1 (4.6)
Statistical Analysis 1: Comparison: Sulforaphane vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.98, Mixed Models Analysis — The test was considered statistically significant if the p-value < 0.05; Mixed-effects model with random intercept and unstructured covariance matrix from baseline to week 16; Mean Difference (Final Values) = 0.08, Standard Error of Mean 2.99 — This analysis compares LS Mean Sulforaphane - LS Mean Placebo

3. Primary Outcome: Social Responsiveness Scale-2 (SRS-2) Total Score at Week 8
Description: as for outcome 1
Time Frame: Week 8
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
T-score | 73.7 (7.4) | 74.5 (4.6)
Statistical Analysis 1: Comparison: Sulforaphane vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.797, Mixed Models Analysis — The test was considered statistically significant if the p-value < 0.05; Mixed-effects model with random intercept and unstructured covariance matrix from baseline to week 16; Mean Difference (Final Values) = -0.774, Standard Error of Mean 2.99 — This analysis compares LS Mean Sulforaphane - LS Mean Placebo

4. Primary Outcome: Social Responsiveness Scale-2 (SRS-2) Total Score at Week 12
Description: as for outcome 1
Time Frame: Week 12
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
T-score | 75.3 (7.4) | 72.9 (4.6)
Statistical Analysis 1: Comparison: Sulforaphane vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.442, Mixed Models Analysis — The test was considered statistically significant if the p-value < 0.05; Mixed-effects model with random intercept and unstructured covariance matrix from baseline to week 16; Mean Difference (Final Values) = 2.32, Standard Error of Mean 3.01 — This analysis compares LS Mean Sulforaphane - LS Mean Placebo

5. Primary Outcome: Social Responsiveness Scale-2 (SRS-2) Total Score at Week 16
Description: as for outcome 1
Time Frame: Week 16
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
T-score | 75.5 (7.4) | 72.7 (4.6)
Statistical Analysis 1: Comparison: Sulforaphane vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.373, Mixed Models Analysis — The test was considered statistically significant if the p-value < 0.05; Mixed-effects model with random intercept and unstructured covariance matrix from baseline to week 16; Mean Difference (Final Values) = 2.72, Standard Error of Mean 3.05 — This analysis compares LS Mean Sulforaphane - LS Mean Placebo

6. Secondary Outcome: Social Responsiveness Scale-2 (SRS-2) Subscale Score (Social Awareness)
Description: The Social Responsiveness Scale-2 (SRS-2) is a 65-item caregiver report that includes 5 subscales covering core symptom domains of ASD (Social Awareness, Social Cognition, Social Communication, Social Motivation, and Restricted Interests/ Repetitive Behaviors). The SRS-2-Social Awareness subscale measures a participant's ability to recognize social cues. This subscale comprises 8 items with scores ranging from 1 to 4 for a total range of scores from 8 to 32. A higher score represents a greater ability to recognize social cues.
  Subscales are not diagnostic in nature, but they provide some insight into individual behaviors. This subscale was measured at Baseline, Week 4, Week 8, Week 12, and Week 16.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
score on a scale
  Baseline | 10.9 (2.5) | 10.9 (1.6)
  Week 4 | 10.5 (2.5) | 11.3 (1.6)
  Week 8 | 10.6 (2.5) | 11.3 (1.6)
  Week 12 | 10.8 (2.5) | 11.0 (1.6)
  Week 16 | 10.7 (2.5) | 11.2 (1.6)

7. Secondary Outcome: Social Responsiveness Scale-2 (SRS-2) Subscale Score (Social Cognition)
Description: The Social Responsiveness Scale-2 (SRS-2) is a 65-item caregiver report that includes 5 subscales covering core symptom domains of ASD (Social Awareness, Social Cognition, Social Communication, Social Motivation, and Restricted Interests/ Repetitive Behaviors). The SRS-2-Social Cognition subscale measures a participant's ability to interpret social behavior. This subscale comprises 12 items with scores ranging from 1 to 4 for a total range of scores from 12 to 48. A higher score represents a greater ability to interpret social behaviors. Subscales are not diagnostic in nature, but they provide some insight into individual behaviors. This subscale was measured at Baseline, Week 4, Week 8, Week 12, and Week 16.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
score on a scale
  Baseline | 19.1 (4.1) | 17.4 (2.6)
  Week 4 | 18.3 (4.1) | 18.2 (2.6)
  Week 8 | 18.2 (4.1) | 18.4 (2.6)
  Week 12 | 18.7 (4.1) | 17.9 (2.6)
  Week 16 | 18.7 (4.1) | 17.9 (2.6)

8. Secondary Outcome: Social Responsiveness Scale-2 (SRS-2) Subscale Score (Social Communication)
Description: The Social Responsiveness Scale-2 (SRS-2) is a 65-item caregiver report that includes 5 subscales covering core symptom domains of ASD (Social Awareness, Social Cognition, Social Communication, Social Motivation, and Restricted Interests/ Repetitive Behaviors). The SRS-2-Social Communication subscale measures a participant's ability to assess reciprocal communication in social situations. This subscale comprises 22 items with scores ranging from 1 to 4 for a total range of scores from 22 to 88. A higher score represents a greater ability to assess reciprocal communication. Subscales are not diagnostic in nature, but they provide some insight into individual behaviors. This subscale was measured at Baseline, Week 4, Week 8, Week 12, and Week 16.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
score on a scale
  Baseline | 34.0 (6.6) | 32.0 (4.1)
  Week 4 | 32.4 (6.6) | 33.6 (4.1)
  Week 8 | 32.6 (6.6) | 33.5 (4.1)
  Week 12 | 34.1 (6.6) | 32.0 (4.1)
  Week 16 | 34.4 (6.6) | 31.7 (4.1)

9. Secondary Outcome: Social Responsiveness Scale-2 (SRS-2) Subscale Score (Social Motivation)
Description: The Social Responsiveness Scale-2 (SRS-2) is a 65-item caregiver report that includes 5 subscales covering core symptom domains of ASD (Social Awareness, Social Cognition, Social Communication, Social Motivation, and Restricted Interests/ Repetitive Behaviors). The SRS-2-Social Motivation subscale measures the degree to which a participant is motivated to participate in social interactions. This subscale comprises 11 items with scores ranging from 1 to 4 for a total range of scores from 11 to 44. A higher score represents a greater motivation to participate in social interaction. Subscales are not diagnostic in nature, but they provide some insight into individual behaviors. This subscale was measured at Baseline, Week 4, Week 8, Week 12, and Week 16.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
score on a scale
  Baseline | 15.5 (4.1) | 14.7 (2.5)
  Week 4 | 14.8 (4.1) | 15.4 (2.5)
  Week 8 | 14.6 (4.1) | 15.6 (2.5)
  Week 12 | 15.5 (4.1) | 14.7 (2.5)
  Week 16 | 15.9 (4.1) | 14.3 (2.5)

10. Secondary Outcome: Social Responsiveness Scale-2 (SRS-2) Subscale Score (Restricted Interests/Repetitive Behaviors)
Description: The Social Responsiveness Scale-2 (SRS-2) is a 65-item caregiver report that includes 5 subscales covering core symptom domains of ASD (Social Awareness, Social Cognition, Social Communication, Social Motivation, and Restricted Interests/ Repetitive Behaviors). The SRS-2-Restricted Interests/Repetitive Behaviors subscale assesses the participant's level of stereotypy and circumscribed interests. This subscale comprises 12 items with scores ranging from 1 to 4 for a total range of scores from 12 to 48. A higher score represents a greater level of stereotypy and circumscribed interests. Subscales are not diagnostic in nature, but they provide some insight into individual behaviors. This subscale was measured at Baseline, Week 4, Week 8, Week 12, and Week 16.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
score on a scale
  Baseline | 18.6 (4.5) | 17.6 (2.8)
  Week 4 | 18.1 (4.5) | 18.2 (2.8)
  Week 8 | 17.7 (4.5) | 18.5 (2.8)
  Week 12 | 18.7 (4.5) | 17.5 (2.8)
  Week 16 | 18.5 (4.5) | 17.7 (2.8)

11. Secondary Outcome: Aberrant Behavior Checklist (ABC) Subscale Score (Social Withdrawal)
Description: The Aberrant Behavior Checklist (ABC) is a 58-item caregiver questionnaire developed to assess medication effects in individuals with developmental disorders and includes 5 distinct subscales of behavioral symptoms. The ABC-Social Withdrawal subscale assesses the participant's level social withdrawal. This subscale comprises 16 items with scores ranging from 0 to 3 for a total range of scores from 0 to 48. A higher score represents a greater level of social withdrawal. This subscale was measured at Baseline, Week 4, Week 8, Week 12, and Week 16.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
score on a scale
  Baseline | 8.7 (5.1) | 8.3 (3.2)
  Week 4 | 8.2 (5.1) | 8.8 (3.2)
  Week 8 | 8.2 (5.1) | 8.8 (3.2)
  Week 12 | 9.0 (5.1) | 8.1 (3.2)
  Week 16 | 9.5 (5.1) | 7.5 (3.2)

12. Secondary Outcome: Aberrant Behavior Checklist (ABC) Subscale Scores (Hyperactivity)
Description: The Aberrant Behavior Checklist (ABC) is a 58-item caregiver questionnaire developed to assess medication effects in individuals with developmental disorders and includes 5 distinct subscales of behavioral symptoms. The ABC-Hyperactivity subscale assesses the participant's level hyperactivity and non-compliance. This subscale comprises 16 items with scores ranging from 0 to 3 for a total range of scores from 0 to 48. A higher score represents a greater level of hyperactivity/non-compliance. This subscale was measured at Baseline, Week 4, Week 8, Week 12, and Week 16.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
score on a scale
  Baseline | 14.3 (5.7) | 10.8 (3.6)
  Week 4 | 13.0 (5.7) | 12.1 (3.6)
  Week 8 | 12.6 (5.7) | 12.5 (3.6)
  Week 12 | 13.7 (5.7) | 11.3 (3.6)
  Week 16 | 13.6 (5.7) | 11.5 (3.6)

13. Secondary Outcome: Aberrant Behavior Checklist (ABC) Subscale Score (Inappropriate Speech)
Description: The Aberrant Behavior Checklist (ABC) is a 58-item caregiver questionnaire developed to assess medication effects in individuals with developmental disorders and includes 5 distinct subscales of behavioral symptoms. The ABC-Inappropriate Speech subscale assesses the participant's use of inappropriate speech. This subscale comprises 4 items with scores ranging from 0 to 3 for a total range of scores from 0 to 12. A higher score represents a greater use of inappropriate speech. This subscale was measured at Baseline, Week 4, Week 8, Week 12, and Week 16.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
score on a scale
  Baseline | 3.4 (1.7) | 2.8 (1.1)
  Week 4 | 3.2 (1.7) | 2.9 (1.1)
  Week 8 | 3.0 (1.7) | 3.1 (1.1)
  Week 12 | 3.3 (1.7) | 2.9 (1.1)
  Week 16 | 3.5 (1.7) | 2.6 (1.1)

14. Secondary Outcome: Aberrant Behavior Checklist (ABC) Subscale Score (Stereotypy)
Description: The Aberrant Behavior Checklist (ABC) is a 58-item caregiver questionnaire developed to assess medication effects in individuals with developmental disorders and includes 5 distinct subscales of behavioral symptoms. The ABC-Stereotypy subscale assesses the participant's level of stereotypic behavior. This subscale comprises 7 items with scores ranging from 0 to 3 for a total range of scores from 0 to 21. A higher score represents a greater level of stereotypic behavior. This subscale was measured at Baseline, Week 4, Week 8, Week 12, and Week 16.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
score on a scale
  Baseline | 1.3 (3.2) | 2.2 (2.0)
  Week 4 | 1.1 (3.2) | 2.4 (2.0)
  Week 8 | 1.0 (3.2) | 2.5 (2.0)
  Week 12 | 1.3 (3.2) | 2.2 (2.0)
  Week 16 | 1.6 (3.2) | 1.6 (2.0)

15. Secondary Outcome: Aberrant Behavior Checklist (ABC) Subscale Score (Irritability)
Description: The Aberrant Behavior Checklist (ABC) is a 58-item caregiver questionnaire developed to assess medication effects in individuals with developmental disorders and includes 5 distinct subscales of behavioral symptoms. The ABC-Irritability subscale assesses the participant's level of irritability. This subscale comprises 15 items with scores ranging from 0 to 3 for a total range of scores from 0 to 45. A higher score represents a greater level of irritability. This subscale was measured at Baseline, Week 4, Week 8, Week 12, and Week 16.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
score on a scale
  Baseline | 9.6 (5.1) | 8.3 (3.2)
  Week 4 | 9.4 (5.1) | 8.6 (3.2)
  Week 8 | 9.7 (5.1) | 8.3 (3.2)
  Week 12 | 9.7 (5.1) | 8.3 (3.2)
  Week 16 | 9.8 (5.1) | 8.1 (3.2)

16. Secondary Outcome: Clinical Global Impression-Severity (CGI-S) Score
Description: The CGI-Severity (CGI-S) scale is a 7-point, clinician-rated scale providing an overall assessment of patient functioning relative to other patients with a similar diagnosis (1=not at all ill to 7=severely ill). A higher score indicates a higher level of severity of psychopathology. This scale was measured at Baseline, Week 4, Week 8, Week 12, and Week 16.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
units on a scale
  Baseline | 4.74 (0.6) | 4.56 (0.3)
  Week 4 | 4.70 (0.6) | 4.60 (0.3)
  Week 8 | 4.71 (0.6) | 4.58 (0.3)
  Week 12 | 4.72 (0.6) | 4.58 (0.3)
  Week 16 | 4.70 (0.6) | 4.60 (0.3)

17. Secondary Outcome: Number of Participants With Clinical Global Impression-Improvement (CGI-I) Score of Much Improved or Very Much Improved
Description: The clinician-rated CGI-Improvement (CGI-I) scale rates overall improvement or worsening of illness (ie, ASD) relative to baseline. The CGI-Improvement (CGI-I) scale rates overall improvement or worsening of illness (ie, ASD) relative to baseline. Possible scores on this scale range from 1-6 with the following assigned values: 1 = "Very Much Improved"; 2 = "Much Improved; 3 = "Minimally improved"; 4 = "No change"; 5 = "Minimally worse"; 6= "Much worse." A higher score indicates worsening of illness (ie, ASD), whereas a lower score indicates improvement of illness. This scale was measured at Week 4, Week 8, Week 12, and Week 16. In this measure, the number of participants in each treatment arm determined by the study physician to be "Much Improved" or "Very Much Improved" (indicative of meaningful clinical improvement) were counted.
Time Frame: Week 4, Week 8, Week 12, Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
Participants
  Week 4: Very Much Improved or Much Improved | 3 | 1
  Week 4: No Improvement to Very Much Worse | 21 | 23
  Week 8: Very Much Improved or Much Improved | 4 | 2
  Week 8: No Improvement to Very Much Worse | 20 | 22
  Week 12: Very Much Improved or Much Improved | 3 | 4
  Week 12: No Improvement to Very Much Worse | 21 | 20
  Week 16: Very Much Improved or Much Improved | 0 | 1
  Week 16: No Improvement to Very Much Worse | 24 | 23

18. Secondary Outcome: Repetitive Behavior Scale-Revised (RBSR) Total Score
Description: The RBS-R is a 43-item, informant-based questionnaire designed to quantify a range of restricted, repetitive behaviors (RRB) observed in ASD. Scores for each item range from 0 = "Behavior does not occur" to 3 = "Behavior occurs and is a severe problem". Thus the total range is 0 to 129. A higher score indicates a higher breadth of repetitive behaviors. This scale was measured at Baseline, Week 4, Week 8, Week 12, and Week 16.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
score on a scale
  Baseline | 23.0 (14.0) | 22.3 (8.7)
  Week 4 | 21.7 (14.0) | 23.5 (8.7)
  Week 8 | 23.3 (14.0) | 22.0 (8.7)
  Week 12 | 23.3 (14.0) | 22.0 (8.7)
  Week 16 | 24.2 (14.0) | 21.0 (8.7)

19. Secondary Outcome: Mean Red Blood Cell Value
Description: This measure assesses the red blood cell value as part of the complete blood count measurement. This blood count measure was assessed at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: 10^6 cells/microliter
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
10^6 cells/microliter
  Baseline | 5.0 (0.3) | 5.1 (0.3)
  Week 12 | 5.1 (0.3) | 5.0 (0.3)

20. Secondary Outcome: Mean White Blood Cell Value
Description: This measure assesses the white blood cell value as part of the complete blood count measurement. This blood count measure was assessed at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: 10^3 cells/microliter
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
10^3 cells/microliter
  Baseline | 6.3 (2.3) | 6.5 (2.2)
  Week 12 | 6.0 (1.8) | 6.9 (2.2)

21. Secondary Outcome: Mean Hemoglobin Value
Description: This measure assesses the hemoglobin value as part of the complete blood count measurement. This blood count measure was assessed at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
g/dL
  Baseline | 14.8 (1.4) | 15.0 (1.1)
  Week 12 | 15.0 (1.2) | 14.5 (1.0)

22. Secondary Outcome: Mean Hematocrit Value
Description: This measure assesses the hematocrit value as part of the complete blood count measurement. This blood count measure was assessed at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: percentage of volume of whole blood
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
percentage of volume of whole blood
  Baseline | 43.8 (3.5) | 44.4 (2.9)
  Week 12 | 44.4 (3.0) | 43.2 (2.8)

23. Secondary Outcome: Mean Corpuscular Volume Value
Description: This measure assesses the mean corpuscular volume value as part of the complete blood count measurement. This blood count measure was assessed at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: femtoliter
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
femtoliter
  Baseline | 87.3 (3.2) | 86.8 (4.6)
  Week 12 | 87.8 (3.1) | 86.6 (3.8)

24. Secondary Outcome: Mean Corpuscular Hemoglobin Value
Description: This measure assesses the mean corpuscular hemoglobin value as part of the complete blood count measurement. This blood count measure was assessed at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: picogram
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
picogram
  Baseline | 29.4 (1.7) | 29.3 (1.8)
  Week 12 | 29.7 (1.2) | 29.2 (1.8)

25. Secondary Outcome: Mean Corpuscular Hemoglobin Concentration Value
Description: This measure assesses the mean corpuscular hemoglobin concentration value as part of the complete blood count measurement. This blood count measure was assessed at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
g/dL
  Baseline | 33.8 (1.0) | 33.9 (1.1)
  Week 12 | 33.8 (0.9) | 33.7 (0.9)

26. Secondary Outcome: Mean Red Blood Cell Distribution Width Value
Description: This measure assesses the red blood cell distribution width value as part of the complete blood count measurement. This blood count measure was assessed at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: % of volume of whole blood
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
% of volume of whole blood
  Baseline | 13.6 (0.8) | 13.7 (1.0)
  Week 12 | 13.6 (0.9) | 13.6 (1.0)

27. Secondary Outcome: Mean Platelets Value
Description: This measure assesses the platelets value as part of the complete blood count measurement. This blood count measure was assessed at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: 10^3 cells/microliter
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
10^3 cells/microliter
  Baseline | 253.8 (74.7) | 286.0 (67.5)
  Week 12 | 246.0 (69.5) | 279.3 (57.7)

28. Secondary Outcome: Mean Absolute Neutrophils Value
Description: This measure assesses the absolute neutrophils value as part of the complete blood count measurement. This blood count measure was assessed at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: 10^3 cells/microliter
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
10^3 cells/microliter
  Baseline | 3.5 (2.0) | 3.7 (1.8)
  Week 12 | 3.3 (1.5) | 6.3 (11.0)

29. Secondary Outcome: Mean Absolute Lymphocytes Value
Description: This measure assesses the absolute lymphocytes value as part of the complete blood count measurement. This blood count measure was assessed at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: 10^3 cells/microliter
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
10^3 cells/microliter
  Baseline | 2.1 (0.6) | 2.1 (0.5)
  Week 12 | 1.9 (0.6) | 3.5 (6.9)

30. Secondary Outcome: Mean Absolute Monocytes Value
Description: This measure assesses the absolute monocytes value as part of the complete blood count measurement. This blood count measure was assessed at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: 10^3 cells/microliter
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
10^3 cells/microliter
  Baseline | 0.5 (0.2) | 0.6 (0.2)
  Week 12 | 0.5 (0.1) | 0.9 (1.6)

31. Secondary Outcome: Mean Absolute Eosinophils Value
Description: This measure assesses the absolute eosinophils value as part of the complete blood count measurement. This blood count measure was assessed at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: 10^6 cells/microliter
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
10^6 cells/microliter
  Baseline | 0.2 (0.1) | 0.1 (0.1)
  Week 12 | 0.2 (0.1) | 0.2 (0.2)

32. Secondary Outcome: Mean Absolute Basophils Value
Description: This measure assesses the absolute basophils value as part of the complete blood count measurement. This blood count measure was assessed at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: 10^3 cells/microliter
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
10^3 cells/microliter
  Baseline | 0.013 (0.034) | 0.013 (0.034)
  Week 12 | 0.004 (0.021) | 0.009 (0.029)

33. Secondary Outcome: Mean Serum Chemistries (Sodium)
Description: This measure assesses the change in the patient's sodium levels. This serum chemistry level was measured at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: millimol/liter
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
millimol/liter
  Baseline | 140.6 (2.3) | 141.0 (2.0)
  Week 12 | 141.8 (2.5) | 141.3 (1.8)

34. Secondary Outcome: Mean Serum Chemistries (Potassium)
Description: This measure assesses the change in the patient's potassium levels. This serum chemistry level was measured at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
mmol/L
  Baseline | 4.4 (0.4) | 4.5 (0.4)
  Week 12 | 4.7 (0.6) | 4.5 (0.4)

35. Secondary Outcome: Mean Serum Chemistries (Chloride)
Description: This measure assesses the change in the patient's chloride levels. This serum chemistry level was measured at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
mmol/L
  Baseline | 100.1 (2.1) | 99.6 (1.9)
  Week 12 | 100.1 (2.3) | 100.7 (2.1)

36. Secondary Outcome: Mean Serum Chemistries (Bicarbonate)
Description: This measure assesses the change in the patient's bicarbonate levels. This serum chemistry level was measured at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
mmol/L
  Baseline | 22.8 (3.0) | 22.3 (1.5)
  Week 12 | 23.1 (2.7) | 22.8 (2.4)

37. Secondary Outcome: Mean Serum Chemistries (Blood Urea Nitrogen)
Description: This measure assesses the change in the patient's blood urea nitrogen levels. This serum chemistry level was measured at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
mg/dL
  Baseline | 13.0 (4.8) | 11.4 (2.8)
  Week 12 | 13.3 (4.3) | 11.6 (3.5)

38. Secondary Outcome: Mean Serum Chemistries (Creatinine)
Description: This measure assesses the change in the patient's creatinine levels. This serum chemistry level was measured at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
mg/dL
  Baseline | 0.8 (0.1) | 0.8 (0.2)
  Week 12 | 0.8 (0.1) | 0.8 (0.2)

39. Secondary Outcome: Mean Serum Chemistries (Glucose)
Description: This measure assesses the change in the patient's glucose levels. This serum chemistry level was measured at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
mg/dL
  Baseline | 90.9 (13.0) | 91.1 (12.6)
  Week 12 | 87.0 (18.3) | 86.3 (13.5)

40. Secondary Outcome: Mean Liver Function Tests Values (Alanine Transaminase)
Description: This measure assesses the change in the patient's level of liver function through measure of alanine transaminase (ALT). This liver function test value was measured at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
IU/L
  Baseline | 22.1 (16.7) | 26.0 (18.0)
  Week 12 | 29.6 (40.7) | 20.7 (10.8)

41. Secondary Outcome: Mean Liver Function Tests Values (Aspartate Transaminase)
Description: This measure assesses the change in the patient's level of liver function through measure of aspartate transaminase. This liver function test value was measured at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
IU/L
  Baseline | 22.3 (10.2) | 21.9 (5.8)
  Week 12 | 25.2 (10.6) | 19.8 (5.1)

42. Secondary Outcome: Mean Liver Function Tests Values (Total Bilirubin)
Description: This measure assesses the change in the patient's level of liver function through measure of total bilirubin. This liver function test value was measured at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
mg/dL
  Baseline | 0.5 (0.3) | 0.4 (0.3)
  Week 12 | 0.5 (0.2) | 0.5 (0.4)

43. Secondary Outcome: Mean Value of Thyroid Stimulating Hormone (TSH)
Description: This measure assesses the change in the patient's value of thyroid stimulating hormone. This hormone value was measured at Baseline and Week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: milli-international units/ microliter
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
milli-international units/ microliter
  Baseline | 2.3 (1.2) | 2.2 (1.2)
  Week 12 | 2.3 (1.2) | 1.8 (1.1)

44. Secondary Outcome: Least Squares Mean of Vital Signs (Weight)
Description: This measure assesses the change in the patient's weight (lbs). This vital sign was measured at Baseline, Week 4, Week 8, Week 12, and Week 16.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Measure: Least Squares Mean (Standard Error); unit: pounds
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
pounds
  Baseline | 147.1 (28.1) | 148.3 (17.4)
  Week 4 | 147.2 (28.1) | 148.2 (17.4)
  Week 8 | 146.8 (28.1) | 148.6 (17.4)
  Week 12 | 146.9 (28.1) | 148.6 (17.4)
  Week 16 | 146.8 (28.1) | 148.6 (17.4)

45. Secondary Outcome: Least Squares Mean of Vital Signs (Height)
Description: This measure assesses the change in the patient's height (centimeters). This vital sign was measured at Baseline, Week 4, Week 8, Week 12, and Week 16.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Measure: Least Squares Mean (Standard Error); unit: centimeters
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
centimeters
  Baseline | 173.9 (6.5) | 173.3 (4.0)
  Week 4 | 173.9 (6.5) | 173.3 (4.0)
  Week 8 | 173.9 (6.5) | 173.3 (4.0)
  Week 12 | 173.9 (6.5) | 173.3 (4.0)
  Week 16 | 173.9 (6.5) | 173.3 (4.0)

46. Secondary Outcome: Least Squares Mean of Vital Signs (Blood Pressure)
Description: This measure assesses the change in the patient's systolic and diastolic blood pressure. This vital sign was measured at Baseline, Week 4, Week 8, Week 12, and Week 16.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
mmHg
  Baseline Systolic | 115.2 (6.6) | 116.7 (4.1)
  Baseline Diastolic | 69.8 (4.5) | 70.6 (2.8)
  Week 4 Systolic | 116.3 (6.6) | 115.5 (4.1)
  Week 4 Diastolic | 69.7 (4.5) | 70.7 (2.8)
  Week 8 Systolic | 116.4 (6.6) | 115.4 (4.1)
  Week 8 Diastolic | 69.6 (4.5) | 70.8 (2.8)
  Week 12 Systolic | 116.2 (6.6) | 115.7 (4.1)
  Week 12 Diastolic | 71.0 (4.5) | 69.4 (2.8)
  Week 16 Systolic | 116.2 (6.6) | 115.7 (4.1)
  Week 16 Diastolic | 71.1 (4.5) | 69.3 (2.8)

47. Secondary Outcome: Least Squares Mean of Vital Signs (Heart Rate)
Description: This measure assesses the change in the patient's heart rate (beats per minute). This vital sign was measured at Baseline, Week 4, Week 8, Week 12, and Week 16.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Measure: Least Squares Mean (Standard Error); unit: Beats per Minute
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 24 | 24
Beats per Minute
  Baseline | 86.1 (8.6) | 87.5 (5.4)
  Week 4 | 88.0 (8.6) | 85.6 (5.4)
  Week 8 | 87.8 (8.6) | 85.7 (5.4)
  Week 12 | 86.5 (8.6) | 87.0 (5.4)
  Week 16 | 90.0 (8.6) | 83.5 (5.4)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from baseline to week 16 (a total of 16 weeks).
Description: Adverse conditions were collected prior to randomization and allocation of treatment at baseline. Participants who described any of these symptoms as worsening (or becoming present) over the 16 weeks of the study were classified as having an adverse event.
Arm/Group | Sulforaphane | Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 14/24 | 14/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sulforaphane (N=24) | Placebo (N=24)
Aggression (Psychiatric disorders) | 2 | 2
Anxiety (Psychiatric disorders) | 1 | 0
Appetite Decrease (Gastrointestinal disorders) | 0 | 1
Difficulty Falling Asleep (Psychiatric disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Irritability (Psychiatric disorders) | 3 | 4
Localized Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 2 | 1
Sedation (Psychiatric disorders) | 0 | 1
Self-injurious Behavior (Psychiatric disorders) | 0 | 2
Stereotypy (Psychiatric disorders) | 1 | 1
Stomach Discomfort (Gastrointestinal disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/59/NCT02909959/Prot_SAP_000.pdf